CLINICAL TRIAL: NCT01780090
Title: Handheld Technology for Speech Development in Students With Autism Spectrum Disorders (ASDs)
Brief Title: Handheld Technology for Speech Development in Students With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Handhold Adaptive (Other)
Responsible Party: Principal Investigator, Frederick Shic, Assistant Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1208010627; ED-IES-12-R-0007 (Other Grant/Funding Number: Department of Education)
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Autism Spectrum Disorders
Keywords: autism; prosody; speech; autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Speech

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iPad software (Experimental): Student participants will use specialized, iPad software under the direction of the SLP, 1 time a week over the course of 2 months.
  Interventions: Other: iPad software

INTERVENTIONS:
Other: iPad software — A specialized iPad application, entitled SpeechPrompts, has been developed to treat prosodic difficulties commonly seen in ASDs. SpeechPrompts provides the SLPs that work with students with ASDs an additional tool to treat prosody. The SpeechPrompts software offers visual support and biofeedback to change prosody. These two tools are not typically available for school-based SLPs.

SUMMARY:
The proposed study will result in a software application compatible with the Apple iPad, iPhone and iPod Touch (hereafter termed "iOS devices") which addresses several aspects of prosodic deficits common in speakers with Autism Spectrum Disorders (ASDs) and other communication disorders, using a developmentally appropriate, intuitive interface that requires little technical skill and which can be managed by educators and parents. The program will contain elements that aid in tracking and maintaining individual student progress records, and will be designed for use in the classroom, at home, and in other environments. This study's intended focus is on the feasibility and usability of the software application.

ELIGIBILITY:
Inclusion Criteria:

* SLPs, in Connecticut Public Schools, who provide intervention to students with autism spectrum disorders.
* Students, ages 4 - 19, who attend school in Connecticut and demonstrate prosodic difficulties secondary to a diagnosis of ASD.

Exclusion Criteria:

* Students with concommitant genetic disorders

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Learning of software | 3 months
  Assessment of Outcome:
  Each speech-language pathologist (SLP) will complete a software training then take a post-training online assessment measuring software competency.
Usability of software | 3 months
  Assessment of Outcome:
  SLPs will complete satisfaction surveys and attend a focus group to obtain information regarding software usability.

SECONDARY OUTCOMES:
Student engagement in treatment | 3 months
  Assessment of Outcome:
  SLPs will rate the student's engagement using a rating scale after each treatment session with the iPad and software.
Software effectiveness | 3 months
  Assessment of Outcome:
  SLPs will rate student participants' prosody before and after iPad treatment using a specialized rubric to measure changes in speech production.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Shic, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States